CLINICAL TRIAL: NCT06217146
Title: A Two-part Study, Part I an Open-label; and Part II a Randomized Double-blind, Placebo-controlled Study to Evaluate the Safety and Efficacy of MediCane's Medical Cannabis Oil for Treatment of Agitation and Disruptive Behaviors in Subjects With Dementia Including Probable Alzheimer's Disease (AD)
Brief Title: A Medical Cannabis Oil for Treatment of Agitation and Disruptive Behaviors in Subjects With Dementia.
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Part I: Open-label was completed.
Sponsor: M. H MediCane Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: AGM-01
Record Dates: First submitted 2023-11-20; First posted 2024-01-22 (Actual); Last update posted 2024-06-27 (Actual); Status verified 2024-06

CONDITIONS: Agitation,Psychomotor; Disruptive Behavior; Dementia; Alzheimer Disease
MeSH Terms: conditions — Psychomotor Agitation; Problem Behavior; Dementia; Alzheimer Disease | interventions — Medical Marijuana

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MediCane's medical cannabis oil (Experimental)
  Interventions: Drug: Medical Cannabis
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo Oil

INTERVENTIONS:
Drug: Medical Cannabis — MediCane's medical cannabis oil
  Arms: MediCane's medical cannabis oil
Drug: Placebo Oil — Placebo Oil
  Arms: Placebo

SUMMARY:
This double-blind, placebo-controlled study is designed to assess the effectiveness of, MediCane's medical cannabis oil extracted from MediCane's proprietary strain into GMP-grade olive oil, as an add-on therapy to standard of care (SoC), in reducing agitation and disruptive behaviors in subjects with dementia including probable AD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are Male or Female age ≥50 years.
* Subjects have a diagnosis of major neurocognitive disorder (previously dementia) according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-V) Criteria for at least 6 months prior to screening or a diagnosis of probable AD using the NINCDS-ADRDA clinical criteria.
* Subjects on antipsychotic medications may be included in the study.
* Subject exhibits agitation/aggression with a Neuropsychiatric Inventory (NPI-12)-agitation/aggression subdomain score of four or higher (≥4) at screening.
* Subject has a legal guardian who is able and willing to provide ICF and able to provide - information in writing. The caregiver should be spending enough time with the subject on a regular basis in order to provide valid information as requested.
* Subjects are on stable SoC for treatment of agitation and disruptive behaviors for at least 2 weeks prior to the screening visit.
* Subjects on Acetyl Choline Esterase inhibitors, antifungals, macrolide antibiotics and anti-hypertensive therapy including ACE inhibitors should be on stable doses for at least 2 weeks prior to screening visit or if changed, at least 2 weeks prior to visit 1.
* Subject's Mini Mental State Exam score (MMSE) is 24 or less at screening.

Exclusion Criteria:

* Subject without a legal guardian.
* Subject with any current unstable medical condition.
* Subject has any unstable condition involving fluid retention, pulmonary infiltrates, congestive heart failure, respiratory symptoms or disease, or cardiac symptoms or disease.
* Subject has one of the following hepatic /renal disorders:

  1. Confirmed and unexplained impaired hepatic function as indicated by screening AST or ALT>3 the upper limit of normal (ULN) or total bilirubin > 2 ULN.
  2. Chronic kidney disease of Stage > 4, according to National Kidney Foundation Kidney Disease Outcome Quality Initiative guidelines for chronic kidney disease.
* Subject has epilepsy.
* Subject has a history of hypersensitivity to any cannabinoid.
* Subject has the presence or history of a primary psychotic psychiatric disorder or subject has clinically significant delusions or hallucinations secondary to the neurodegenerative disease (NPI-12 delusions or hallucinations sub-score of 4 or higher (≥4).
* Subject suffering from delirium as defined in Appendix B - Criteria for Delirium.
* Current inpatient hospitalization.
* Subject has other health-related factors that could explain behavioral disturbances (electrolyte disturbances, infectious diseases, etc.).
* Subject has a satisfactory response to antipsychotic treatments.
* Subjects treated with one of the following medications: opiates, primidone, phenobarbitol, carbamazepine, rifampicin, rifabutin, troglitazone, hypericum perforatum, or valproic acid within 30 days from Visit 1.
* Subjects currently on medication known to interact with Cannabis-based medications are excluded; Subjects taking Cannabis-based therapies are excluded if within the past 2 weeks from Visit 1.
* Subjects with a history of addiction or drug abuse.

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2022-10-12 (Actual); Primary Completion 2024-03-10 (Actual); Study Completion 2024-03-10 (Actual)

PRIMARY OUTCOMES:
Part 1 Safety (Adverse Events) | Up to 22 weeks
  Number of participants with treatment-related adverse events as assessed by severity. protocol.
Part 2 Efficacy (CMAI) | 12 weeks
  Change in agitation and aggression from baseline to Week 12 as measured using the Cohen-Mansfield Agitation Inventory-Community (CMAI-C), a 37-item scale that measures the types and frequencies of agitated behaviors, each rated on a 7-point scale of frequency, where higher scores indicate greater agitation severity.

SECONDARY OUTCOMES:
Part 1 Efficacy (NPI-12) | up to 18 weeks
  Change in neuropsychiatric symptoms measured by the total score and subscores of the NPI-12.

CONTACTS AND LOCATIONS:
Overall Officials: Neta Rimmerman, PhD, Study Director — Sponsor GmbH
Locations (3):
- Israel (3):
  - Laniado Hospital, Netanya
  - Sheba Medical Center, Ramat Gan
  - Tel-Aviv Sourasky Medical Center Ichilov, Tel Aviv

IPD SHARING:
Plan to Share IPD: No